CLINICAL TRIAL: NCT00454090
Title: A Phase I, Open-Label, Multi-centre Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Oral Doses of AZD8330 in Patients With Advanced Malignancies
Brief Title: AZD8330 First Time in Man in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1536C00001
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Cancer
Keywords: Advanced Malignancies
MeSH Terms: conditions — Neoplasms | interventions — AZD8330

INTERVENTIONS:
Drug: AZD8330 — oral tablet
  Other Names: ARRY-424704

SUMMARY:
The primary purpose of this protocol is to investigate the safety and tolerability of AZD8330 (ARRY-424704) in patients with Advanced Malignancies

ELIGIBILITY:
Inclusion Criteria:

* Cancer which is refractory to standard therapies, or no therapies exist;

Exclusion Criteria:

* Participated in radiotherapy, biological or chemotherapy within 21 days prior to study start;
* Hasn't participated in investigation drug study within 30 days;
* Brain metastases/spinal cord compression unless treated and stable,
* Off steroids/anticonvulsants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2007-03; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of AZD8330 in patient with advanced malignancies.
Outcome variables: Adverse Events, Clinical Chemistry, Haematology, Urinalysis, Vital signs, MUGA scans/echocardiography, ECGs, Ophthalmologic examination, O2 saturation

SECONDARY OUTCOMES:
To determine the PK of AZD8330.
To investigate possible PD/PK relationships
To investigate effect of AZD8330 on pERK in PBMCs

CONTACTS AND LOCATIONS:
Overall Officials: Emerging Oncology Medical Science Director, MD, Study Director — AstraZeneca
Locations (3):
- United States (2):
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Houston, Texas
- Research Site, Oslo, Norway

REFERENCES:
- [Derived] Cohen RB, Aamdal S, Nyakas M, Cavallin M, Green D, Learoyd M, Smith I, Kurzrock R. A phase I dose-finding, safety and tolerability study of AZD8330 in patients with advanced malignancies. Eur J Cancer. 2013 May;49(7):1521-9. doi: 10.1016/j.ejca.2013.01.013. Epub 2013 Feb 21. PMID 23433846